CLINICAL TRIAL: NCT03148496
Title: Tissue Reinforcement of Incisional Closure Among High Risk Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic and the halt to elective surgeries hindered enrollment; PI left insitution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Julie Holihan, Assistant Professor of Surgery-Clinical, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-17-0063
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Wound Complication
Keywords: abdominal surgery; wound complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Biologic Mesh and Small Bites (Experimental): Biologic mesh placement and small bites used for suturing.
  Interventions: Device: Biologic Mesh; Procedure: Small Bites
- Small Bites and No Biologic Mesh (Experimental): Small bites used for suturing with no placement of biologic mesh
  Interventions: Procedure: Small Bites
- Biologic mesh and Large Bites (Experimental): Biologic mesh placement and large bites used for suturing
  Interventions: Device: Biologic Mesh; Procedure: Large Bites
- Large Bites and no biologic mesh (Active Comparator): Large bites used for suturing and no placement of biologic mesh.
  Interventions: Procedure: Large Bites

INTERVENTIONS:
Device: Biologic Mesh — Biologic mesh placed during surgery
  Arms: Biologic Mesh and Small Bites; Biologic mesh and Large Bites
Procedure: Small Bites — 0.5 cm x 0.5 cm sutures used
  Arms: Biologic Mesh and Small Bites; Small Bites and No Biologic Mesh
Procedure: Large Bites — 1.0 x 1.0 sutures used
  Arms: Biologic mesh and Large Bites; Large Bites and no biologic mesh

SUMMARY:
Half of all individuals will undergo abdominal surgery in their lifetime. Following abdominal surgery, 30% of patients will suffer a major chronic complication with their wound closure in the first post-operative year. This may include significant wound infections, open wounds, fluid collections, fascial dehiscence, or incisional hernia. These complications not only have a substantial impact on the health care system (cost and chronic disease) and the hospital (cost and space), but most importantly have a substantial impact on the patient. Major chronic wound complications adversely impact patient quality of life and function. Potential methods to reduce major wound complications include utilizing specific suturing techniques or reinforcing the incision line. Suturing technique of small-bites (0.5x0.5 cm bites) as opposed to large bites (1.0x1.0 cm bites) has been shown to be efficacious in European populations with a typical body mass index of 20-25 kg/m2. Tissue reinforcement has been shown to decrease rates of major wound complications in small randomized controlled trials.

However, the lack of widespread adoption of these practices may be due to issues of generalizability including strict inclusion criteria, careful patient selection, and small study size. For example, the generalizability of small bites to an overweight population (mean BMI in the United States is 28 kg/m2) as opposed to a normal-weight population are unclear. The use of synthetic materials in comorbid patients or complex settings may risk major wound complications such as prosthetic infection. Biologic materials have been shown to be effective in decreasing major wound complications but in different settings. This study is being done to assess the effectiveness of different efficacious strategies to decrease the rate of major wound complications following abdominal surgery among high-risk individuals The researchers hypothesize:

1. Among high-risk patients undergoing abdominal surgery, the use of "small-bites" closure as opposed to "large-bites" closure will increase the proportion of patients who are free of major, chronic wound complications at 1-year post-operative.
2. Among high-risk patients undergoing abdominal surgery, the biologic tissue reinforcement of the suture line as opposed to no reinforcement will increase the proportion of patients who are free of major, chronic wound complications at 1-year post-operative.

ELIGIBILITY:
Inclusion Criteria:

All high-risk patients undergoing laparotomy or laparoscopic-assisted abdominal surgery. This includes:

1. all overweight patients (BMI>=25 kg/m2),
2. current smokers,
3. those who are immunosuppressed,
4. those who are malnourished, or
5. those who are undergoing a contaminated case (CDC wound classification of 2 or 3).

Exclusion Criteria:

1. patients unlikely to follow-up in a year (e.g. no phone or lives out of state),
2. patients unlikely to survive more than 2 years based upon surgeon judgment (e.g. metastatic cancer, end-stage cirrhosis),
3. patients where the clinician would not place prosthetic (e.g. pregnant patient, pediatric patient during growth stage),
4. patient has a planned second surgery within the next year (e.g. ostomy reversal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Holihan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon B. Johnson (LBJ) Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodenough CJ, Ko TC, Kao LS, Nguyen MT, Holihan JL, Alawadi Z, Nguyen DH, Flores JR, Arita NT, Roth JS, Liang MK. Development and validation of a risk stratification score for ventral incisional hernia after abdominal surgery: hernia expectation rates in intra-abdominal surgery (the HERNIA Project). J Am Coll Surg. 2015 Apr;220(4):405-13. doi: 10.1016/j.jamcollsurg.2014.12.027. Epub 2015 Jan 2. PMID 25690673
- [Background] Armananzas L, Ruiz-Tovar J, Arroyo A, Garcia-Peche P, Armananzas E, Diez M, Galindo I, Calpena R. Prophylactic mesh vs suture in the closure of the umbilical trocar site after laparoscopic cholecystectomy in high-risk patients for incisional hernia. A randomized clinical trial. J Am Coll Surg. 2014 May;218(5):960-8. doi: 10.1016/j.jamcollsurg.2014.01.049. Epub 2014 Feb 18. PMID 24680572
- [Background] McCarthy M Jr, Jonasson O, Chang CH, Pickard AS, Giobbie-Hurder A, Gibbs J, Edelman P, Fitzgibbons R, Neumayer L. Assessment of patient functional status after surgery. J Am Coll Surg. 2005 Aug;201(2):171-8. doi: 10.1016/j.jamcollsurg.2005.03.035. PMID 16038812
- [Background] Hawn MT, Itani KM, Giobbie-Hurder A, McCarthy M Jr, Jonasson O, Neumayer LA. Patient-reported outcomes after inguinal herniorrhaphy. Surgery. 2006 Aug;140(2):198-205. doi: 10.1016/j.surg.2006.02.003. PMID 16904970
- [Background] Blackstock R, Hernandez NC. Characterization of the macrophage subset affected and its response to a T suppressor factor (TsFmp) found in cryptococcosis. Infect Immun. 1989 Oct;57(10):2931-7. doi: 10.1128/iai.57.10.2931-2937.1989. PMID 2777368
- [Background] Holihan JL, Henchcliffe BE, Mo J, Flores-Gonzalez JR, Ko TC, Kao LS, Liang MK. Is Nonoperative Management Warranted in Ventral Hernia Patients With Comorbidities?: A Case-matched, Prospective, Patient-centered Study. Ann Surg. 2016 Oct;264(4):585-90. doi: 10.1097/SLA.0000000000001865. PMID 27355269
- [Background] Deerenberg EB, Harlaar JJ, Steyerberg EW, Lont HE, van Doorn HC, Heisterkamp J, Wijnhoven BP, Schouten WR, Cense HA, Stockmann HB, Berends FJ, Dijkhuizen FPH, Dwarkasing RS, Jairam AP, van Ramshorst GH, Kleinrensink GJ, Jeekel J, Lange JF. Small bites versus large bites for closure of abdominal midline incisions (STITCH): a double-blind, multicentre, randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1254-1260. doi: 10.1016/S0140-6736(15)60459-7. Epub 2015 Jul 15. PMID 26188742
- [Background] Millbourn D, Cengiz Y, Israelsson LA. Effect of stitch length on wound complications after closure of midline incisions: a randomized controlled trial. Arch Surg. 2009 Nov;144(11):1056-9. doi: 10.1001/archsurg.2009.189. PMID 19917943
- [Background] Millbourn D, Cengiz Y, Israelsson LA. Risk factors for wound complications in midline abdominal incisions related to the size of stitches. Hernia. 2011 Jun;15(3):261-6. doi: 10.1007/s10029-010-0775-8. Epub 2011 Jan 30. PMID 21279664
- [Background] Bhangu A, Fitzgerald JE, Singh P, Battersby N, Marriott P, Pinkney T. Systematic review and meta-analysis of prophylactic mesh placement for prevention of incisional hernia following midline laparotomy. Hernia. 2013 Aug;17(4):445-55. doi: 10.1007/s10029-013-1119-2. Epub 2013 May 28. PMID 23712289
- [Background] Fortelny RH, Hofmann A, May C, Kockerling F; BioMesh Study Group. Prevention of a Parastomal Hernia by Biological Mesh Reinforcement. Front Surg. 2015 Oct 22;2:53. doi: 10.3389/fsurg.2015.00053. eCollection 2015. PMID 26557646
- [Background] Muysoms FE, Detry O, Vierendeels T, Huyghe M, Miserez M, Ruppert M, Tollens T, Defraigne JO, Berrevoet F. Prevention of Incisional Hernias by Prophylactic Mesh-augmented Reinforcement of Midline Laparotomies for Abdominal Aortic Aneurysm Treatment: A Randomized Controlled Trial. Ann Surg. 2016 Apr;263(4):638-45. doi: 10.1097/SLA.0000000000001369. PMID 26943336
- [Background] Sarr MG, Hutcher NE, Snyder S, Hodde J, Carmody B. A prospective, randomized, multicenter trial of Surgisis Gold, a biologic prosthetic, as a sublay reinforcement of the fascial closure after open bariatric surgery. Surgery. 2014 Oct;156(4):902-8. doi: 10.1016/j.surg.2014.06.022. PMID 25239343
- [Background] Bali C, Papakostas J, Georgiou G, Kouvelos G, Avgos S, Arnaoutoglou E, Papadopoulos G, Matsagkas M. A comparative study of sutured versus bovine pericardium mesh abdominal closure after open abdominal aortic aneurysm repair. Hernia. 2015 Apr;19(2):267-71. doi: 10.1007/s10029-014-1262-4. Epub 2014 May 13. PMID 24820007
- [Background] Ferzoco SJ. A systematic review of outcomes following repair of complex ventral incisional hernias with biologic mesh. Int Surg. 2013 Oct-Dec;98(4):399-408. doi: 10.9738/INTSURG-D-12-00002.1. PMID 24229031
- [Background] Stampfer MJ, Buring JE, Willett W, Rosner B, Eberlein K, Hennekens CH. The 2 x 2 factorial design: its application to a randomized trial of aspirin and carotene in U.S. physicians. Stat Med. 1985 Apr-Jun;4(2):111-6. doi: 10.1002/sim.4780040202. PMID 4023472
- [Derived] Coelho R, Dhanani NH, Lyons NB, Bernardi K, Askenasy EP, Millas S, Holihan JL, Ali Z, Liang MK. Hernia Prevention Using Biologic Mesh and/or Small Bites: A Multispecialty 2 x 2 Factorial Randomized Controlled Trial. J Am Coll Surg. 2023 Aug 1;237(2):309-317. doi: 10.1097/XCS.0000000000000705. Epub 2023 Apr 11. PMID 37458369

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 163 participants enrolled, 107 met inclusion criteria and were randomized
Period: Overall Study
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Started | 27 | 28 | 25 | 27
Completed | 20 | 19 | 19 | 26
Not Completed | 7 | 9 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh | Total
Number analyzed (Participants) | 27 | 28 | 25 | 27 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 23 | 20 | 92
  >=65 years | 4 | 2 | 2 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 9 | 13 | 48
  Male | 12 | 17 | 16 | 14 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 23 | 16 | 18 | 76
  Not Hispanic or Latino | 8 | 5 | 9 | 9 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 25 | 27 | 107

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Major Chronic Wound Infection
Description: Proportion of participants with major chronic wound infection
Time Frame: 1 year after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Major Complications
Description: Major complications include surgical site infection, ventral incisional hernia, and/or reoperation
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 27 | 28 | 25 | 27
Participants | 5 | 5 | 6 | 4

3. Secondary Outcome: Number of Participants With Surgical Site Infections
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 27 | 28 | 25 | 27
Participants | 2 | 1 | 1 | 0

4. Secondary Outcome: Number of Participants With Reoperations
Description: any unplanned invasive procedure involving the fascia, mesh, or peritoneal cavity
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 27 | 28 | 25 | 27
Participants | 2 | 1 | 2 | 2

5. Secondary Outcome: Operative Duration
Description: length of the entire procedure
Time Frame: about 119 minutes to 337 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 27 | 28 | 25 | 27
minutes | 210.19 (70.96) | 205.50 (70.96) | 230.64 (106.48) | 180.26 (61.58)

6. Secondary Outcome: Participants Quality of Life as Assessed by Activities Assessment Scale
Description: Quality of life is scored from 1 to 100, where the higher the score the higher quality of life
Time Frame: 1 year after surgery
Population: Data were not collected for 13 participants in the Biologic Mesh arm. Data were not collected for 10 participants in the No Biologic Mesh arm. Data were not collected for 7 participants in the Large Bites arm. Data were not collected for 16 participants in the Small Bites arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Biologic Mesh: Biologic mesh placement
  Biologic Mesh: Biologic mesh placed during surgery
- No Biologic Mesh: No placement of biologic mesh
- Large Bites: large bites used for suturing
  Large Bites: 1.0 x 1.0 sutures used
- Small Bites: Small bites used for suturing
  Small Bites: 0.5 cm x 0.5 cm sutures used
Arm/Group | Biologic Mesh | No Biologic Mesh | Large Bites | Small Bites
Number analyzed (Participants) | 39 | 45 | 45 | 39
score on a scale | 64 (33) | 70 (31) | 68 (32) | 66 (32)

7. Secondary Outcome: Participants Health Status as Assessed by the Euroqol-5D Questionnaire
Description: Health Status is scored from 0 to 100, where the higher the score the better the health
Time Frame: 1 year after surgery
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Biologic Mesh | No Biologic Mesh | Large Bites | Small Bites
Number analyzed (Participants) | 39 | 45 | 45 | 39
score on a scale | 80 [60 to 100] | 80 [60 to 100] | 80 [55 to 100] | 80 [70 to 100]

8. Secondary Outcome: Cost Analyses
Description: calculated from the hospital's perspective by assessing charges for all patient visits, admissions, and procedures
Time Frame: 1 year after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Surgeon Perception
Description: likert type and open ended questions assessing perception, barriers and likelihood of utilizing interventions outside of the trial
Time Frame: 1 year after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Major Complications
Description: Major complications include surgical site infection, ventral incisional hernia, and/or reoperation
Time Frame: 3 years after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Surgical Site Infections
Time Frame: 3 years after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Reoperations
Description: any unplanned invasive procedure involving the fascia, mesh, or peritoneal cavity
Time Frame: 3 years after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Participants Quality of Life as Assessed by Activities Assessment Scale
Description: Quality of life is scored from 1 to 100, where the higher the score the higher quality of life
Time Frame: 3 years after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh | No Biologic Mesh | Large Bites | Small Bites
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Participants Health Status as Assessed by the Euroqol-5D Questionnaire
Description: Health Status is scored from 0 to 100, where the higher the score the better the health
Time Frame: 3 years after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh | No Biologic Mesh | Large Bites | Small Bites
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Cost Analyses
Description: calculated from the hospital's perspective by assessing charges for all patient visits, admissions, and procedures
Time Frame: 3 years after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Surgeon Perception
Description: as for outcome 9
Time Frame: 3 years after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year post surgery
Arm/Group | Biologic Mesh and Small Bites | Small Bites and No Biologic Mesh | Biologic Mesh and Large Bites | Large Bites and no Biologic Mesh
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28 | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/27 | 1/28 | 2/25 | 2/27
Other Adverse Events (participants affected / at risk) | 4/27 | 5/28 | 5/25 | 2/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biologic Mesh and Small Bites (N=27) | Small Bites and No Biologic Mesh (N=28) | Biologic Mesh and Large Bites (N=25) | Large Bites and no Biologic Mesh (N=27)
Reoperation (Surgical and medical procedures) | 2 | 1 | 2 | 2
Bowel Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biologic Mesh and Small Bites (N=27) | Small Bites and No Biologic Mesh (N=28) | Biologic Mesh and Large Bites (N=25) | Large Bites and no Biologic Mesh (N=27)
Ventral incisional hernia (General disorders) | 2 | 4 | 4 | 2
Surgical Site Infection (Infections and infestations) | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03148496/Prot_SAP_000.pdf